CLINICAL TRIAL: NCT02212327
Title: Testing Tissue Sodium Stores in Continuous Ambulatory Peritoneal Dialysis (CAPD) Patients Receiving Icodextrin or Glucose-Based Dialysate, A Randomized Trial-Aims 1 & 2
Brief Title: Testing Tissue Sodium Stores in CAPD Patients-Aims 1 & 2
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Alp Ikizler, Professor, Vanderbilt University Medical Center
Other Study IDs: 140157
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: End Stage Renal Disease
Keywords: Na+ MRI; salt stores
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood and urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PD subjects
- Controls

SUMMARY:
The investigators' overarching goal is to improve long-term outcomes for end stage renal disease (ESRD) patients. In this study we focus specifically on patients receiving peritoneal dialysis (PD). Volume regulation in PD patients is related to hypertension, heart failure, nutritional status, and survival. Salt (NaCl) is the body's ion transport target to normally regulate volume via the kidneys; however, in hemodialysis (HD) patients the dialyser or in PD patients the peritoneal membrane, must serve that purpose. Determining volume status in PD patients is not easy and monitoring sodium (Na+) is more difficult still. The investigators have developed a novel, noninvasive approach to this problem involving 23Na+ magnetic resonance imaging (Na-MRI). Na+ is stored bound to proteoglycans in mostly the skin. Our technique measures Na+ in skin and skeletal muscle. In this study, we propose to apply this novel technique to PD patients.

Aim 1. To determine Na+ stores in PD patients, to compare Na+ stores to normal controls using Na-MRI technique, and to correlate Na+ stores by Na-MRI with multifrequency bioimpedance measurements and cross-sectional clinical data.

Hypothesis: Na+ stores are increased in PD patients compared to normal controls; they are increased in PD patients with volume expansion and in those patients with high soluble vascular endothelial growth factor receptor-3 (sFlt-4) levels.

Aim 2. To determine the utility of Na-MRI as an assessment of preserving residual renal function in PD patients.

Hypothesis: Extracellular volume expansion as measured by multifrequency bioimpedance was found to have no utility in predicting preservation of residual renal function in PD patients. The investigators hypothesize that Na+ stores as determined by 23Na-MRI will fulfill that function and will be inversely, rather than directly, related.

ELIGIBILITY:
Inclusion Criteria:

Both subject groups:

* Age 18 to 80 years;
* BMI < 40;
* Ability to give informed consent;
* Life expectancy greater than 6 months.

PD subjects:

* On peritoneal dialysis for greater than 3 months;
* Using glucose lactate-buffered PD solutions with consistent glucose exposure;
* Stable peritoneal prescription (Kt/V > 1.7 or Tccr > 50 ml/week/1.73 m2).

Control subjects:

* Estimated glomerular filtration rate (GFR) ≥ 60 ml/min/1.73m2;
* No proteinuria.

Exclusion Criteria (both subject groups):

* Pregnancy;
* Intolerance to study protocols;
* Severe, unstable, active, or chronic inflammatory disease (congestive heart failure-NY Class IV, active infection, active connective tissue disorder, active cancer or cancer history in the prior 5 years, HIV, liver disease, including active chronic hepatitis B or C);
* Active inflammatory conditions [systemic lupus erythematosus (SLE), rheumatoid arthritis (RA), minimal change disease (MCD)];
* Patients prescribed or being treated with spironolactone;
* History of cirrhosis;
* Poor compliance with dialysis prescription.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients on PD and healthy controls
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2014-08; Primary Completion 2016-11-29 (Actual); Study Completion 2016-11-29 (Actual)

PRIMARY OUTCOMES:
Aim 1: Na+ stores in PD subjects vs. controls | baseline
Aim 2: a change in Na+ stores in PD subjects | baseline and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alp Ikizler, MD, Principal Investigator — Vanderbilt University; Jens Titze, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States